CLINICAL TRIAL: NCT00501839
Title: How Long Should First-line Treatment be Continued in Infertile PCOS Patients Who Ovulate Under Clomiphene Citrate? A Randomized Controlled Clinical Study.
Brief Title: Clomiphene Citrate in Infertile PCOS Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2006a
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: Anovulation; Clomiphene citrate; Infertility; PCOS; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Anovulation | interventions — Clomiphene

ARMS (3):
- Group A (Active Comparator): Cyclic progestogens for nine months
  Interventions: Drug: clomiphene citrate
- Group B (Active Comparator): CC treatment for further three cycles at the same ovulating doses followed by six months of cyclic progestogens
  Interventions: Drug: clomiphene citrate
- Group C (Active Comparator): CC administration at the same ovulating doses for nine cycles
  Interventions: Drug: clomiphene citrate

INTERVENTIONS:
Drug: clomiphene citrate

SUMMARY:
Anovulatory infertility is a common feature of the polycystic ovary syndrome (PCOS). Clomiphene citrate (CC) represents the first therapeutic option for treating the anovulatory infertility in PCOS patients because it is characterized by low costs, limited dose-dependent side effects, and simplicity of administration and management due to no need for ongoing monitoring.

Excellent results in terms of ovulations have been obtained using CC. However, only 50% of patients who ovulates under CC will conceive. The exact explanation for the discrepancy between the ovulation and pregnancy rates is unknown, but several hypotheses on the anti-estrogenic effects that CC exerts on the ovary and uterus have been suggested.

To date, few data are available on the optimal schedule for CC administration, and it is unknown how long patients who ovulate under CC should continue treatment before switching to second-line ovulation induction therapy. The aim of the study was to define the clinical benefits of CC administration according to its duration of administration.

DETAILED DESCRIPTION:
Infertile PCOS patients who had three previous ovulatory cycles under CC will be enrolled and randomized in three groups (groups A, B, and C). In group A, patients will receive cyclic progestogens for nine months; in group B, patients will continue CC treatment for further three cycles at the same ovulating doses followed by six months of cyclic progestogens; and in group C, patients will continue CC administration at the same ovulating doses for nine cycles. In each case, CC will be administered using a traditional incremental-doses protocol up to 150 mg daily.

All patients eligible will undergo baseline assessment consisting of anthropometric, hormonal, and ultrasonographic evaluations. During the study, the clinical and reproductive outcomes, and the adverse experience will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant. Continuous variables will be analyzed with the unpaired t test and general linear model for repeated measures analysis with Bonferroni test for the post-hoc analysis as required. For categorical variables, the Pearson chi-square and Fisher's exact tests will be used. Cumulative pregnancy rate, our primary end-point, will be calculated by the Kaplan-Maier method, and the differences between the two groups will be assessed with the log-rank test. Cox proportional-hazards model will be used to calculate the hazard ratio for new pregnancy in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using NIH criteria)
* Anovulatory infertility (using WHO criteria)
* Previous three CC-stimulated ovulatory cycles

Exclusion Criteria:

* Age <18 or >35 years
* Severe obesity (BMI >35)
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugs
* Intention to start a diet or a specific program of physical activity
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cumulative pregnancy rate | 12 months

SECONDARY OUTCOMES:
Ovulation rate Abortion rate Live-birth rate Adverse events Multiple pregnancy rate | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Magna Graecia" of Catanzaro; Francesco Orio, MD, Principal Investigator — Department of Endocrinology, University "Federico II" of Naples; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Federico II" of Naples
Locations (1):
- Pugliese Hospital, Catanzaro, Catanzaro, CZ, Italy, Italy

REFERENCES:
- [Background] Palomba S, Orio F Jr, Falbo A, Russo T, Tolino A, Zullo F. Clomiphene citrate versus metformin as first-line approach for the treatment of anovulation in infertile patients with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Sep;92(9):3498-503. doi: 10.1210/jc.2007-1009. Epub 2007 Jun 26. PMID 17595241
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746